CLINICAL TRIAL: NCT00965822
Title: A Randomized, Double-blind, Placebo-controlled Study on the Efficacy and Safety of CVT-E002 in the Treatment of Upper Respiratory Tract Infections in a Pediatric (3-11 Years) Population
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Afexa Life Sciences Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CVT-E002-2007-3
Record Dates: First submitted 2009-08-25; First posted 2009-08-26 (Estimated); Last update posted 2012-08-31 (Estimated); Status verified 2012-08

CONDITIONS: Upper Respiratory Tract Infections
Keywords: URTI; Natural Health Products
MeSH Terms: conditions — Respiratory Tract Infections | interventions — COLD-fX

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator)
  Interventions: Other: North American ginseng
- 2 (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Other: North American ginseng — 3 day, once daily, dosing
  Other Names: COLD-FX
  Arms: 1
Other: Placebo — 3 day, once daily dosing
  Arms: 2

SUMMARY:
Parents with children aged 3-11 will participate in this study. About 500 children will take part in the study. We expect about half of those children will develop symptoms of a respiratory infection. Active participation in this study will last 14 days after a parent reports symptoms of a respiratory infection in a participant. Those children who do meet the study criteria of symptoms will then be randomly placed (like a flip of a coin) into one of 2 groups to take either COLD-FX® or placebo for 3 days. A placebo will look exactly like COLD-FX® but contains no active ingredients. The participant has an equal chance of being placed in either of the above groups. The study is double-blind, so neither the participant nor the study staff will know which study group the participant was placed in until the study is completed. If this information is needed in an emergency at any time throughout the study, it is quickly available from the sponsor.

Participation in the study will be for 14 days after symptoms of a respiratory infection are reported to study staff. Your child will take the study product for 3 days, you will complete a daily diary, receive 4 phone calls and be seen for a final study visit to review the diary and complete a final health check of your child.

DETAILED DESCRIPTION:
The primary objective is to assess the efficacy of acute dosing of CVT-E002 in reducing the duration of URTI symptoms in children 3-11 years of age.

The secondary objectives are to asses the efficacy of acute dosing of CVT-E002 in reducing: (1) symptom severity; (2) peak CARIFS scores and; (3) absenteeism for participant and/or parent/guardian. The ease of administration and the safety of acute dosing of CVT-E002 in children 3-11 years of age will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy individuals of both genders aged years 3 - 11
2. Willing to adhere to the requirements of the protocol, including availability for follow-up visits
3. Parent/guardian willing and able to sign written consent

Exclusion Criteria:

1. Medical conditions:

   * Asthma requiring treatment in the last 3 months with oral steroids - prednisone greater than 10 mg/day
   * Received influenza vaccination for the winter season when the trial is run.
   * Active tuberculosis
   * Cystic fibrosis
   * Significant pulmonary disorders (chronic bronchitis, emphysema or other chronic respiratory illness)
   * Any ongoing allergen immunotherapy during study or for 6 months prior HIV/AIDS
   * Malignancy (under active observation or treatment)
   * Unstable cardiovascular disease (physician visit or hospitalization for unstable cardiovascular disease in the last 6 months)
   * Known renal abnormalities (serum creatinine known to be > upper limit for age group)
   * Acute or active chronic liver disease
   * Diabetes
   * Neurological or psychiatric disease (progressive or currently under treatment)
   * Bleeding disorders
   * Major surgery in the last 6 months or planned surgery over the course of the study
   * Crohn's disease, Juvenile arthritis, Ulcerative Colitis or any other autoimmune disease
   * Other serious medical conditions
2. Medications:

   * Medications for allergic rhinitis/conjunctivitis, including: antihistamines; oral, parenteral, nasal, and ophthalmic corticosteroids; cromolyn sodium; nedocromil; and intranasal anticholinergics (If the participants agree to stop taking these products prior to study entry and for the duration of the study, they can participate in the study.)
   * Oral or long-acting beta-agonists, theophylline, and leukotriene modifiers
   * Phenelzine
   * Pentobarbital
   * Haloperidol
   * Warfarin
   * Heparin
   * Immunosuppressants

     * Any other natural health products or dietary supplements, with the exception of vitamins and minerals with dose of <600 mg/day of vitamin E and containing no vitamin K. Natural health products or dietary supplements include products such as, but not limited to, Echinacea, Ginseng (beverages, foods, extracts, capsules, or tablets), St. John's Wort, Gingko, Glucosamine, Fish Oil supplements, Evening Primrose Oil, Green Tea or other herbal products consumed in the form of a pill or capsule. (If the participants agree to stop taking these products prior to study entry and for the duration of the study, they can participate in the study.)
3. Known allergy to any ingredient in the study product or placebo, including: ginseng, icing sugar, stevia leaf powder, mixed berries natural flavour (MC010946), grape natural flavour (MC010947) or caramel color liquid (DN700 caramelan 8-110).

Ages: 3 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 293 (Actual)
Dates: Start 2009-09; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
The primary objective is to assess the efficacy of acute dosing of CVT-E002 in reducing the duration of URTI symptoms in children 3-11 years of age | 14 days

SECONDARY OUTCOMES:
To asses the efficacy of acute dosing of CVT-E002 in reducing: (1) symptom severity; (2) peak CARIFS scores and; (3) absenteeism for participant and/or parent/guardian. | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Shelly McNeil, FRCPC, Principal Investigator — Dalhousie University
Locations (4):
- Canada (4):
  - Alberta Health Services, Edmonton, Alberta
  - Saint John Regional Hospital, Saint John, New Brunswick
  - Canadian Center for Vaccinology, Dalhousie University, Halifax, Nova Scotia
  - JDM Research, Toronto, Ontario